CLINICAL TRIAL: NCT06937333
Title: Investigation of Pain, Cervical Joint Range of Motion, and Sleep Quality in Children With Bruxism
Brief Title: Pain and Mobility in Children With Sleep Bruxism
Status: Completed | Type: Observational
Sponsor: Karabuk University (Other)
Responsible Party: Principal Investigator, METEHAN YANA, Director, PT, PhD, Karabuk University
Other Study IDs: Karabuk-007
Record Dates: First submitted 2025-04-10; First posted 2025-04-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Bruxism, Sleep
MeSH Terms: conditions — Sleep Bruxism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sleep bruxism: Children diagnosed with sleep bruxism were included in this study.
- Control Group: Age- and sex-matched healthy children were included.

SUMMARY:
Bruxism is defined as a repetitive jaw muscle activity characterized by clenching and grinding teeth caused by mandibular movement. Sleep bruxism is frequently seen and can affect the quality of life of individuals. Since bruxism is characterized by clenching teeth, it can cause pain. However, the relationship between bruxism and pain has not been sufficiently studied in the literature. The relationship between the temporamandibular joint and the cervical region is known. However, the relationship between bruxism and cervical mobility is not clear. Since there may be temporamandibular joint problems in bruxism, it can affect joint movement. The sleep quality of individuals may decrease and this may lead to problems in functionality. However, when the literature is examined, the relationship between bruxism and functional independence in children has not been explained. Therefore, the aim of the study was to compare the pain, range of motion, sleep quality and functional independence of children with bruxism and healthy controls.

DETAILED DESCRIPTION:
Bruxism is defined as repetitive jaw muscle activity characterized by clenching and grinding teeth caused by mandibular movement. Sleep bruxism is frequently seen and can affect the quality of life of individuals. Since bruxism is characterized by clenching teeth, it can cause pain. However, the relationship between bruxism and pain has not been sufficiently studied in the literature. In addition, bruxism can cause problems in joint mobility of the cervical region by affecting the activation of muscles. Although the relationship between the temporomandibular joint and the cervical region is clearly known, the relationship between bruxism and cervical mobility is not clear. For this reason, sleep problems are frequently seen in individuals. The sleep quality of individuals decreases and can cause problems in functionality. However, when the literature is examined, the relationship between bruxism and functional independence in children has not been explained. Since bruxism can reduce the quality of life of individuals due to the indirect effects it causes, it should be seen and evaluated not only as a disorder involving the jaw joint, but as a problem affecting the entire body. Therefore, the aim of the study was to compare pain, range of motion, sleep quality and functional independence in children with bruxism and healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with Nocturnal Bruxism
* Having received parental consent to participate in the study
* Being between the ages of 13-18
* Being in good mental condition
* Being able to understand and follow the instructions in the study
* Having Class 1 occlusion

Exclusion Criteria:

* Not consenting to participate in the study or withdrawing from the study
* Not being able to cooperate well
* Having a history of surgery
* Having any physical disability or chronic disease
* Having received dental treatment in the last 6 months

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children with bruxism and healthy controls
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2024-06-15 (Actual); Primary Completion 2025-02-15 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Pain pressure threshold | Baseline
  Pain pressure threshold was evaluated the algometer.
Range of motion | Baseline
  Cervical range of motion was evaluated with the cervical range of motion device (CROM) developed by the University of Minnesota, USA,
Functional Independence | Baseline
  Functional Independence was evaluated the with the Pediatric Functional Independence Measure. The total score varies between 18-126 and as the score increases, the dependency increases.
Sleep quality | Baseline
  Sleep quality was evaluated the Pitsburg Sleep Quality Index. The total score ranges from 0 to 21, and as the score increases, sleep quality decreases.

CONTACTS AND LOCATIONS:
Overall Officials: Metehan Yana, PhD, Study Director — Karabuk University
Locations (1):
- Karabük University, Karabük, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Brancher LC, Cademartori MG, Jansen K, da Silva RA, Bach S, Reyes A, Boscato N, Goettems ML. Social, emotional, and behavioral problems and parent-reported sleep bruxism in schoolchildren. J Am Dent Assoc. 2020 May;151(5):327-333. doi: 10.1016/j.adaj.2020.01.025. Epub 2020 Mar 26. PMID 32223910